CLINICAL TRIAL: NCT07062237
Title: A Double-Blinded Prospective Randomized Clinical Trial Comparing Euploidy Rates Among Embryos Created From Sibling Oocytes Exposed to Sperm After Ultrashort Abstinence Compared With Standard Abstinence
Brief Title: A Randomized Clinical Trial Comparing Embryo Euploidy Rates Following Ultrashort Versus Standard Abstinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: The Center for Advanced Reproductive Services, P.C. (Other)
Responsible Party: Principal Investigator, Lawrence Engmann, M.D., M.R.C.O.G, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-238-1
Record Dates: First submitted 2025-06-28; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Infertility; Male Factor Infertility
Keywords: Ultrashort abstinence; Sibling oocyte; In vitro fertilization; Euploid embryos
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Sibling oocyte study: Participants will have their oocytes (eggs) divided into two groups. Half of the eggs will be exposed to sperm produced after standard abstinence, and half will be exposed to sperm produced after ultrashort abstinence.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, clinical providers, investigators and outcome assessors will be blinded to outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrashort abstinence (Experimental): Half of participants eggs will be exposed to sperm produced after ultrashort abstinence (1 hour of abstinence).
  Interventions: Other: Ultrashort abstinence
- Standard abstinence (Active Comparator): Half of participants eggs will be exposed to sperm produced after standard abstinence (2-5 days of abstinence).
  Interventions: Other: Standard abstinence

INTERVENTIONS:
Other: Ultrashort abstinence — Ultrashort abstinence: producing a sperm sample after 1 hour of abstinence.
  Arms: Ultrashort abstinence
Other: Standard abstinence — Standard abstinence: producing a sperm sample after 2-5 days of abstinence.
  Arms: Standard abstinence

SUMMARY:
This research is being done to determine if producing sperm after an ultrashort period of abstinence (1 hour of abstinence) will be effective in improving the rates of embryos with normal chromosomes (structures that carry genetic information) during in vitro fertilization (IVF) treatment. The investigators hypothesize that a shorter period of abstinence is effective at improving rates of normal chromosomes among embryos.

DETAILED DESCRIPTION:
As part of the in vitro fertilization (IVF) process, eggs are removed from the ovaries and are inseminated (mixed) or injected with sperm. Typically, sperm samples for IVF are produced on the day of egg retrieval. The current recommendation for abstinence prior to providing this sample is 2-7 days. However, new research has shown that there may be improved IVF outcomes with a shorter period of abstinence including improved integrity of sperm DNA (called sperm DNA fragmentation), sperm parameters (such as motility and shape), embryo quality, implantation rates, pregnancy rates, and live birth rates. One small study found that shorter abstinence may even lead to a higher rate of chromosomally normal embryos.

The purpose of this research study is to determine whether using an ultrashort period of abstinence increases the rates of embryos with normal chromosomes. On the day of egg retrieval, participants will produce two semen samples. The first sample will be collected after 2-5 days of abstinence (standard abstinence). The second sample will be collected 1 hour after the first sample (ultrashort abstinence). Both of these samples will be used for IVF.

At the time of egg retrieval, participants will have their eggs randomized (like the flip of a coin) into two groups. Half of the eggs will be exposed to sperm produced after 2-5 days of abstinence (standard abstinence). The other half of the eggs will be exposed to sperm produced after 1 hour of abstinence (ultrashort abstinence). The goal is to determine the rate of embryos with normal chromosomes in each group. Other goals include looking at how many patients get pregnant after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are nonpregnant females ≥ 18 years and ≤ 42 years of age.
* Subjects obtain greater than or equal to 6 mature oocytes at the time of oocyte retrieval for ICSI or greater than or equal to 8 oocytes at the time of oocyte retrieval for standard insemination.
* Subjects are utilizing standard insemination or ICSI for fertilization.
* Subjects are undergoing PGT-A (PGT for aneuploidy) or PGT-M (PGT for monogenic disorders).
* Subjects are willing to comply with study protocol and procedures and provide written informed consent.

Exclusion Criteria:

* Subjects are utilizing donor oocytes, donor sperm, or gestational carrier.
* Subjects have a diagnosis of cryptozoospermia (no spermatozoa identified in fresh semen sample).
* Subjects are utilizing surgically removed sperm (e.g. via testicular sperm aspiration [TESA] or microsurgical epididymal sperm aspiration [MESA]).
* Subjects are utilizing frozen/thawed sperm, including in cases in which a fresh sample was planned and the sample is insufficient for use.
* Subjects are utilizing frozen/thawed oocytes.
* Subjects undergoing PGT-SR (PGT for structural rearrangements).
* Subjects are undergoing a day 3 (cleavage stage) embryo transfer.
* Subjects obtain less than 6 mature oocytes at the time of oocyte retrieval for ICSI or less than 8 oocytes at the time of oocyte retrieval for standard insemination.
* Subjects obtain greater than or equal to 6 mature oocytes at the time of oocyte retrieval for ICSI or greater than or equal to 8 oocytes at the time of oocyte retrieval for standard insemination but choose to fertilize fewer than 6 (for ICSI) or 8 (for standard insemination).
* Male partner is unable to produce a second semen sample within three hours of the first semen sample (standard abstinence sample)
* Male partner has an infectious disease.

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Non-pregnant females undergoing in vitro fertilization (IVF) with preimplantation genetic testing (PGT) with male partners who can produce a sperm sample
Enrollment: 187 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Euploidy rate per oocyte | Within 2-4 weeks of IVF cycle
  Rate of embryos with normal chromosomes in both groups

SECONDARY OUTCOMES:
Pregnancy rates after transfer of euploid embryos | Within 1-2 weeks of transfer
  Pregnancy rate after one euploid embryo (from either experimental or control group) is transferred back into the participant in a subsequent cycle
Fertilization rate | Within 1 - 2 weeks of IVF cycle
  Proportion of oocytes fertilized in each group
Blastulation rate | Within 2-3 weeks of IVF cycle
  Proportion of usable blastocysts in each group

OTHER OUTCOMES:
Sperm DNA fragmentation and DNA methylation results | 1-2 years after initial study completed
  Compare sperm DNA fragmentation and DNA methylation results between groups

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Advanced Reproductive Services, P.C., Farmington, Connecticut, United States